CLINICAL TRIAL: NCT02169986
Title: Family Practice Resident Research Project: Do Electronic Reminders Increase Adherence of Moisturizer Utilization in Paediatric Atopic Dermatitis?
Brief Title: Atopic Dermatitis Adherence Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-02932
Record Dates: First submitted 2014-04-01; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Atopic Dermatitis/Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- control group (No Intervention): Parents/caregivers will receive the standard of care.
- electronic reminders (Experimental): In this group, the parents/caregivers will receive two daily electronic reminders in addition to the standard of care.
  Interventions: Behavioral: electronic reminders

INTERVENTIONS:
Behavioral: electronic reminders
  Arms: electronic reminders

SUMMARY:
Forgetting is usually listed as the most important cause of low adherence among patients. Most studies to date have looked at the adherence of adults or adolescent population. No studies have been done looking specifically at adherence to topical treatment by parents/caregivers of young children. Our project will try to replicate the same results among the parents/caregivers responsible for children ten years and under. The population in this study will be the parents/caregivers of children 10 and under with atopic dermatitis and the intervention will be the effect of electronic reminders in adherence rates for the use of a moisturizer which is recognized as part of the standard of care in the treatment of atopic dermatitis.

DETAILED DESCRIPTION:
Non Adherence to treatment is a common concern among physicians because it is associated with negative impact on patients' health. Among the different factors that can explain why treatment adherence is so low, forgetfulness is the most common.

Several interventions have been put into practice. Some of them have been proven to be successful, others not. An effective intervention not only has to be successful but also practical.

Technology is an integral part of our everyday lives. In Canada, most adults have access to smartphones, which opens the door to a world of new innovations. Among these are useful applications designed to improve different aspects of every day life.

Electronic reminders are applications designed to send messages, which could improve the adherence to treatment. So far, there are several studies that have proven this benefit in older children and adult population. At this moment, there are no studies involving younger children. Therefore, in this study, the null hypothesis is that electronic reminders will improve the adherence to twice daily application of moisturizers among parents/caregivers of children 10 and under with atopic dermatitis.

The study population will be parents/caregivers of children age 10 and under with atopic dermatitis recruited from Dr. Bergman's paediatric dermatology clinic.

The parents/caregivers of the patients will be invited to participate in this project by the Medical Office Assistant who will send them a letter with the invitation one week before their scheduled appointment. If they agree to participate, they will be asked to sign a consent form and then they will be asked to select an unmarked envelope from a container. The envelopes contain the information for two different groups, one is the experimental and the other the control group.

The experimental group will have the extra task of downloading and utilizing an application called MediSafe. This application will be set up to send reminders two times per day. The control group will be encouraged to continue with the standard of care with no added intervention. Both groups will received a free unlabeled bottle of CeraVe cream. The moisturizer will be unlabeled so as not to allow parents/caregivers perceptions on a specific brand to affect their utilization. External forces such as advertising the parents/caregivers sees or cost of the product could affect the parents/caregivers perception of value and in turn affect adherence.

The parents/caregivers will also receive a calendar in which they have to mark every time their children have moisturizer applied. The calendar will be provided as label on the bottle of moisturizer.

If during the study period the parents/caregivers run out of moisturizer, they can return to the clinic to pick up extra bottles of moisturizer at no cost.

The atopic dermatitis of patients from both groups will be assessed using the EASI score at the beginning and at the end of the 28 days.

Additionally, the parents/caregivers of both groups will be asked to fill up a brief survey form. They will submit this form, along with the calendar label, in an unmarked envelope to maintain anonymity.

The bottles of moisturizer will be weighed before and after the study and also every time a refill of moisturizer is required, to determine the amount of moisturizer used by each group.

This study will follow the standard of care for treatment of atopic dermatitis; no treatment will be withheld.

The principal outcome of this study is to probe whether or not electronic reminders can improve the adherence of moisturizer use in parents/caregivers of children 10 years and under with atopic dermatitis. The changes in the EASI score of the patients after the study and the differences in the amount of moisturizer used per body surface area will be secondary outcomes.

The number of times the calendar label will be marked will reflect the adherence to the treatment. Other data such as severity of eczema, and amount of moisturizer used will be collected. The height, weight, severity of eczema and use of steroid/calcineurin inhibitors will provide additional information that could be used indirectly to measure adherence.

Regarding the data analysis:

Mean differences between the experimental and control groups on adherence and EASI scores will be analyzed using Student's t-test for independent groups. Possible difference on treatment compliance between baseline and post-implementation within the groups will be explored using Student's dependent t-test for paired samples. This pilot study's sample size will be sufficient for the planned analyses, and to help determine effect size and power needed to conduct a larger study on this topic. Univariate descriptive statistics will be reported for all variables.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers of children age 10 and under with atopic dermatitis from Dr. Bergman's dermatology clinic.
* The parents/caregivers must have a smartphone and not already be using an electronic reminder system.
* At least one of the parents/caregivers must have an adequate level of English proficiency in order to follow the instructions required by this project mostly because the electronic reminders are available in English only.

Exclusion Criteria:

* All parents/caregivers of children over the age of 10 with atopic dermatitis.
* Patients receiving systemic immunosuppressive therapy.
* Patients who have a documented sensitivity to CeraVe.
* Parents/caregivers unable to follow instructions in English,
* Parents/caregivers without smartphones.
* Parents/caregivers already using electronic reminders.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Adherence | Effects of electronic reminders on the adherence of 20 parents/caregivers at the end of 28 days study
  The results on adherence of the 20 parents/caregivers in the experimental arm(using electronic reminders) will be contrasted with another 20 parents/caregivers in the control arm.

SECONDARY OUTCOMES:
EASI score changes | The EASI score of the patients' eczema will be measured at the beginning and end of the 28 days study
  The differences in the EASI score on both groups can be used as and indirect measurement of the adherence of the parents/caregivers to the treatment.
Moisturizer | The use of moisturizer among both groups could be used as an indirect measure of adherence to treatment
  The moisturizer jar will be weighted at the beginning and end of the study. That way the amount of moisturizer will be calculated in grams. Because the body surface of the patients in both groups will be obtained at the beginning of the study, the amount of moisturizer per surface can be estimated. If there are significant differences in the use of moisturizer among both groups per unit of surface, this could be used as an indirect measurement of adherence.

CONTACTS AND LOCATIONS:
Overall Officials: James H Bergman, MD, Principal Investigator — University of British Columbia
Locations (1):
- Dr Bergman's Paediatric Dermatologic Clinic, Vancouver, British Columbia, Canada